CLINICAL TRIAL: NCT01729416
Title: Prospective Randomized Controlled Trial Comparing Water Exchange Colonoscopy and Air Colonoscopy in a Community Based Setting
Brief Title: Prospective Randomized Controlled Trial Comparing Water and Air Colonoscopy in a Community Based Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 297959; 297959-4 (Other: UC Davis)
Record Dates: First submitted 2012-11-02; First posted 2012-11-20 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Tubular Adenoma; Colon Cancer; Hyperplastic Polyp
Keywords: colon; cancer; screening; water exchange; air; method; polyp; adenoma; detection; rate; sedation; time; procedure
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms; Polyps; Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water Exchange Colonoscopy (Experimental): The intervention will be water exchange colonoscopy in patients who are randomized to have screening colonoscopy with water exchange colonoscopy.
  Interventions: Other: Water Exchange Colonoscopy
- Air colonoscopy (Active Comparator): The intervention will be colonoscopy using the traditional air method in patients who are randomized to have screening colonoscopy with air colonoscopy.
  Interventions: Other: Air Colonoscopy

INTERVENTIONS:
Other: Water Exchange Colonoscopy — We will turn off the air pump. The colonoscope will be inserted into the rectum and gently advanced. We will suction air pockets as scope is advanced towards the cecum. Water will be infused when encountering closed up lumen. All the infused water will be suctioned out. We will use all other techniques used with conventional air method as needed. For example abdominal pressure, shortening of scope to reduce looping, change of patient position etc.
  We will turn on air pump once cecum reached, or if unsuccessful with water method to open up a close lumen or to go past a tight turn.
  On withdrawal we will continue air insufflation as needed, and closely examine for polyps and remove all visualized polyps. If there is any residual fluid, it will be suctioned out as the scope is withdrawn.
  Arms: Water Exchange Colonoscopy
Other: Air Colonoscopy — Air will be infused into the colon during colonoscopy.
  Arms: Air colonoscopy

SUMMARY:
The purpose of this study is to determine if screening colonoscopy performed on adults with the water exchange method, as opposed to the air method, will have a higher adenoma detection rate.

DETAILED DESCRIPTION:
Screening colonoscopy with removal of pre-cancerous adenomas was recently shown to result in a 53% reduction in mortality from colon cancer. While this clearly validates the practice of screening colonoscopy, missed adenomas, especially in the proximal colon, defined as including cecum, ascending colon, and transverse colon, remains a concern. This was demonstrated in a study of 183 patients who underwent back-to-back colonoscopies. In this population the overall miss rate for adenomas was 24% with proximal adenomas missed more often (27%) than left colon adenomas (21%). Another study looked at 4192 patients in the SEER (Surveillance, Epidemiology, and End Results) Medicare database who developed "interval cancers", that is colon cancer in a patient who had a colonoscopy done in the previous 6-36 months. These interval cancers were predominantly in the proximal colon (Proximal 68%, Distal 19.5%, rectum 10.4%, and unspecified 2.1%). This also suggests that pre-cancerous lesions are being missed in the proximal colon. As such a method that can increase proximal adenoma detection rate would be a welcome change.

One such emerging technique which shows promise for improving adenoma detection rate is water colonoscopy. In one of the early studies employing the water method a trend towards a higher ADR in the water method group was recognized (37% vs. 26%). The observation prompted a retrospective analysis of 1178 cases of screening and surveillance colonoscopy performed by a single endoscopist at the Sacramento VAMC, which showed an overall ADR (presence of at least one adenoma) of 27% with air colonoscopy whereas that for the water method colonoscopy was 35% (p=0.007). In a subsequent combined analysis of two prospective RCT of air vs. water colonoscopy for screening and surveillance using scheduled unsedated colonoscopy [5] and on-demand sedation [6], more patients were found to have at least one diminutive adenoma in the proximal colon in the water method group than in the air group (28% vs. 14%, respectively, p=0.0298). Another quasi randomized study of screening patients performed at Phoenix VAMC using high definition equipment confirmed a significantly higher overall ADR with the water method (n=177) compared with the air method (n=191) (57% vs. 46%) (p=0.03). The odds of detecting an adenoma was 81% higher with the water method (OR 1.81; 95% CI: 1.12-2.90) and independent of age, body mass index (BMI), current smoking and alcohol use, withdrawal time & quality of bowel preparation. In the proximal colon ADR was significantly higher in patients examined with the water method than with air method (46% vs. 35%) (p=0.03), particularly for adenomas <10 mm in size (38% vs. 25%) (p=007). These encouraging preliminary data reflect the potential benefits of water method colonoscopy.

Our current research question is whether this benefit is seen in a community based population as opposed to the VA population which is mostly male and Caucasian.

The investigators plan to perform a prospective, randomized controlled trial comparing proximal adenoma detection rate between a water exchange colonoscopy group and an air colonoscopy group. The investigators intend to employ scheduled sedation, instead of on-demand sedation, to continue the current protocol in place at our institution.

Patients in both the study arms will undergo a split bowel preparation before colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years
* Individuals able to provide informed consent
* Individuals presenting for average-risk colorectal cancer screening by colonoscopy
* Individuals presenting for surveillance of adenomatous/sessile serrated colon polyps as per the US multi-society taskforce on colorectal cancer

Exclusion Criteria:

* Patients who decline to participate
* Prior partial or complete colectomy
* Patients with history of inflammatory bowel disease (ulcerative colitis or Crohn's disease)
* Patients with prior history of colorectal cancer
* Patients with history of screening colonoscopy within the past 10 years
* Patients with history of familial polyposis syndromes (Familial Adenomatous Polyposis, Lynch Syndrome)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Proximal Adenoma detection | Data collected when pathology is available, typically 3-10 days after the patient's procedure. Data is collected only once per patient.
  Presence of adenoma detected anywhere between the cecum and the splenic flexure

SECONDARY OUTCOMES:
Total adenoma detection | Data collected when pathology is available, typically 3-10 days after the patient's procedure. Data is only collected once per patient.
  Adenoma detection anywhere in the colon during colonoscopy.
Sedation requirements | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
  The amount of sedation required to complete the patient's colonoscopy.
Total procedure time | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
  The total time it takes to complete colonoscopy.
Cecal intubation time | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
  The time it takes to reach the cecum during colonoscopy.
Patient position change during procedure | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
  The need for patient's position to be changed from left lateral to other positions, to enable advancement of the colonoscope forward.
Use of colonoscope stiffener during procedure | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
  The need to stiffen the colonoscope to enable to forward movement of the scope during procedure
Abdominal pressure by assistant during procedure | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
  Need for abdominal pressure by endoscopist's assistant during procedure to enable forward movement of colonoscope.
Length of colonoscope at time of cecal intubation | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
  Assessment of length of the colonoscope inserted into the colon to reach the cecum.
Procedure-related pain score | Data collected during and post procedure after recovery from sedation, which is usually within 1 hour post procedure
  Assessment of discomfort due to the procedure, as possible during procedure, and post procedure after recovery from sedation, being cognizant of limitations posed by sedation and attendant amnesia.
Reason for air insufflation, and length of colon when air insufflation started, while performing water colonoscopy | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
  Assessment of percentage of patient requiring air insufflation when water colon fails to open colonic lumen, and site of colon where this is most likely to happen.
Volume of water used during water colonoscopy | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
  Assessment of volume of water introduced into the colon during procedure.
Patient perception regarding air and water colonoscopy | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length.
  Assessment of patient's perception about the 2 methods of colonoscopy.
Advanced adenoma detection rate | Data collected when pathology is available, typically 3-10 days after the patient's procedure. Data is only collected once per patient
Type of polypectomy (cold biopsy/cold snare/snare cautery/need for submucosal injection/need for clip placement) | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length
Bowel preparation quality by Boston Bowel Prep Scale | This will be collected at the time of their procedure appointment which is expected to be 2 to 3 hours in length
Post procedure recovery time | This will be collected at the time of their procedure appointment which is expected to be 2 to 3 hours in length
Serrated polyp detection rate | This will be collected at the time of their procedure appointment which is expected to be 2 to 3 hours in length
Procedure time- morning versus afternoon | This will be collected at the time of their procedure appointment which is expected to be 2 to 3 hours in length
Body Mass Index (BMI) | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length
Smoking history | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length
Alcohol consumption | This will be collected at their procedure appointment which is expected to be 2 to 3 hours in length

CONTACTS AND LOCATIONS:
Overall Officials: Sooraj Tejaswi, M.D., Principal Investigator — University of California, Davis
Locations (1):
- Elk Grove PCN, University of California, Davis, Elk Grove, California, United States

REFERENCES:
- [Background] Zauber AG, Winawer SJ, O'Brien MJ, Lansdorp-Vogelaar I, van Ballegooijen M, Hankey BF, Shi W, Bond JH, Schapiro M, Panish JF, Stewart ET, Waye JD. Colonoscopic polypectomy and long-term prevention of colorectal-cancer deaths. N Engl J Med. 2012 Feb 23;366(8):687-96. doi: 10.1056/NEJMoa1100370. PMID 22356322
- [Background] Rex DK, Cutler CS, Lemmel GT, Rahmani EY, Clark DW, Helper DJ, Lehman GA, Mark DG. Colonoscopic miss rates of adenomas determined by back-to-back colonoscopies. Gastroenterology. 1997 Jan;112(1):24-8. doi: 10.1016/s0016-5085(97)70214-2. PMID 8978338
- [Background] Leung FW, Aharonian HS, Leung JW, Guth PH, Jackson G. Impact of a novel water method on scheduled unsedated colonoscopy in U.S. veterans. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):546-50. doi: 10.1016/j.gie.2008.08.014. PMID 19231497
- [Background] Leung JW, Do LD, Siao-Salera RM, Ngo C, Parikh DA, Mann SK, Leung FW. Retrospective analysis showing the water method increased adenoma detection rate - a hypothesis generating observation. J Interv Gastroenterol. 2011 Jan;1(1):3-7. doi: 10.4161/jig.1.1.14585. PMID 21686105
- [Background] Leung FW, Harker JO, Jackson G, Okamoto KE, Behbahani OM, Jamgotchian NJ, Aharonian HS, Guth PH, Mann SK, Leung JW. A proof-of-principle, prospective, randomized, controlled trial demonstrating improved outcomes in scheduled unsedated colonoscopy by the water method. Gastrointest Endosc. 2010 Oct;72(4):693-700. doi: 10.1016/j.gie.2010.05.020. Epub 2010 Jul 8. PMID 20619405
- [Background] Leung J, Mann S, Siao-Salera R, Ransibrahmanakul K, Lim B, Canete W, Samson L, Gutierrez R, Leung FW. A randomized, controlled trial to confirm the beneficial effects of the water method on U.S. veterans undergoing colonoscopy with the option of on-demand sedation. Gastrointest Endosc. 2011 Jan;73(1):103-10. doi: 10.1016/j.gie.2010.09.020. PMID 21184876
- [Background] Leung FW, Leung JW, Siao-Salera RM, Mann SK. The water method significantly enhances proximal diminutive adenoma detection rate in unsedated patients. J Interv Gastroenterol. 2011 Jan;1(1):8-13. doi: 10.4161/jig.1.1.14587. PMID 21686106
- [Background] Ramirez FC, Leung FW. A head-to-head comparison of the water vs. air method in patients undergoing screening colonoscopy. J Interv Gastroenterol. 2011 Jul;1(3):130-135. doi: 10.4161/jig.1.3.18512. Epub 2011 Jul 1. PMID 22163084
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102